CLINICAL TRIAL: NCT01884311
Title: A Phase III, Multicenter, Open-Label Study to Evaluate the Pharmacokinetics and Safety of Subgam-VF in Primary Immunodeficiency Diseases
Brief Title: Pharmacokinetics (PK) and Safety of Subgam-VF in Primary Immunodeficiency Diseases
Acronym: SCIG03
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCIG03
Record Dates: First submitted 2013-06-14; First posted 2013-06-24 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Primary Immune Deficiency Disorders; Common Variable Immunodeficiency; X-linked Agammaglobulinaemia; Hyperimmunoglobulin M Syndrome
Keywords: Primary Immune Deficiency Disorders; Common Variable Immunodeficiency; X-linked agammaglobulinaemia; Hyper-IgM Syndrome; Subcutaneous; Immunoglobulins
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Common Variable Immunodeficiency; Bruton type agammaglobulinemia; Hyper-IgM Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subgam-VF (Experimental): Subgam-VF is a 16% IgG and will be administered weekly, by subcutaneous infusion. The total duration of treatment will be for 26 weeks.
  Interventions: Biological: Subgam

INTERVENTIONS:
Biological: Subgam — Subgam-VF dose will be given as 1.37 of the established IGIV dose (expressed in mg/kg/week) for 26 weeks (26 infusions) beginning one week after the last IGIV infusion. Dose of Subgam-VF will then be adjusted based on the ratio of the Immunoglobulin G (IgG) average concentration achieved with Subgam-VF compared to IGIV.
  Other Names: Subgam-VF

SUMMARY:
The main objective of the study is to determine the pharmacokinetics profile of Subgam-VF. The secondary objectives are to assess the safety of Subgam-VF and refine the dose adjustment coefficient for Subgam-VF needed for subjects switching from prior intravenous immunoglobulin (IGIV) therapy.

DETAILED DESCRIPTION:
This will be a Phase III, multicenter, open-label, non-randomized study.

Following a screening period, eligible subjects will commence weekly Subgam-VF treatment; this is a 16% subcutaneous IgG product.

Subjects will receive Subgam-VF for 26 weeks during which time safety will be assessed.

After Week 21, PK sampling will commence.

Follow-up visit (one week after the last Subgam-VF infusion, Week 27). All AEs will be monitored up to 28 days after the last Subgam-VF infusion by telephone contact (Week 30).

Subgam-VF will be administered subcutaneously using infusion pumps.

Subjects will be given diaries to record adverse event data as well as any infusions administered at home. In addition there will be a telephone follow up by an appropriately qualified site staff member on day 3 after each site administered and home administered infusion to check for any adverse reactions including infusion site reactions and remind subjects to document these in their subject study diary.

ELIGIBILITY:
Inclusion criteria:

1. Aged between 2 and 75 years (at time of initial consent).
2. Body Mass Index (BMI) < 46 for adults (aged 16 years & older), & BMI < 28 for children.
3. Diagnosed with primary immunodeficiency disease e.g. common variable immunodeficiency, X-linked & autosomal forms of agammaglobulinaemia, hyper-IgM syndrome, Wiskott-Aldrich syndrome.
4. Currently receiving a licensed (or investigational stage III, IIIb) IGIV or SCIG and

   1. IGIV dose is between 300 and 800 mg/kg/month. SCIG dose is between 110 & 300 mg/kg/week;
   2. Dose is stable for at least the past three months (i.e. consistent mg/kg +/- 5%);
   3. The infusion interval is every 21 or 28 days for IGIV & seven days for SCIG;
   4. Has a documented trough level of ≥ 6 g/L (600 mg/dL) on current IgG therapy. If not available can be obtained at the screening visit, Visit 1 (Week 0).
5. Female subjects who are (or become) sexually active must practice contraception by using a method of proven reliability for the duration of the study.
6. Females of child-bearing potential, (defined from the onset of menstruation to one year post menopause), must have a negative result on a urine HCG-based pregnancy test.
7. Willing to comply with all aspects of the protocol, including blood sampling, for the duration of the study.
8. Signed an informed consent form. In the case of subjects under the legal age the parent/guardian will sign an informed consent form & where appropriate the subject will sign an assent form.

Exclusion Criteria:

1. Has a history of any severe anaphylactic reaction to blood or any blood-derived product.
2. Has selective IgA deficiency or has a history of antibodies to IgA.
3. Has clinically significant impairment of cellular or innate immunity at the discretion of the Investigator
4. Has evidence of an active infection at the time of enrolment (i.e. on day of first infusion). Subjects who are asymptomatic but have not completed their course of antibiotics are eligible.
5. Has previously completed or withdrawn from this study.
6. Is currently receiving, or has received, any investigational agent within the prior three months, unless it is an investigational stage III, IIIb IGIV or SCIG.
7. Is pregnant (confirmed by a positive result on an HCG-based pregnancy test) or is nursing.
8. Is positive for any of the following at screening:

   • Serological test for HIV 1&2, HCV, or HBsAg
9. Has levels at screening greater than 2.5 times the upper limit of normal as defined at the central laboratory of any of the following:

   * Alanine transaminase (ALT)
   * Aspartate transaminase (AST)
10. Has severe renal impairment (defined as serum creatinine greater than two times the upper limit of normal or BUN greater than two times the upper limit of normal for the range of the laboratory doing the analysis); the subject is on dialysis; or has a history of acute renal failure.
11. Is known to abuse alcohol, opiates, psychotropic agents, or other chemicals or drugs, or has done so within the past 12 months.
12. Has a history of DVT, or thrombotic complications of IgG therapy, or a prior diagnosis of thrombophilia.
13. Suffers from any acute or chronic medical condition, (e.g. renal disease or predisposing conditions for renal disease, coronary artery disease, or protein losing state, proteinuria) that the Investigator feels may interfere with the conduct of the study.
14. Has an acquired medical condition, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (ANC < 1 x 109/L).
15. Is receiving the following medication:

    * Steroids (long-term daily, > 0.15 mg of prednisone equivalent/kg/day). Requirement for short or intermittent courses of > 0.15mg/kg/day would not exclude a subject.
    * Immunosuppressive drugs
    * Immunomodulatory drugs
16. If ≥ 18 years of age, has non-controlled arterial hypertension (systolic blood pressure > 160 mmHg &/or diastolic blood pressure > 100 mmHg). For younger subjects refer to current guidelines for diagnosis of blood pressure1.
17. Has anemia (hemoglobin < 10 g/dL) at screening.
18. Has severe dermatitis that would preclude sites for safe product administration.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wolford, Study Director — Bio Products Laboratory Limited
Locations (16):
- United States (16):
  - Arizona Allergy Associates, Chandler, Arizona
  - University of California, Irvine, Irvine, California
  - University of California San Diego-- Rady's Children's Hospital, San Diego, California
  - Immunoe International Research, Centennial, Colorado
  - Allergy Associate of the Palm Beaches, North Palm Beach, Florida
  - Ann and Robert H Lurie Children's Hospital, Chicago, Illinois
  - Cardinal Glennon Children's Medical Center, Minneapolis, Minnesota
  - Optimed Research, Columbus, Ohio
  - Oklahoma Institute of Allergy & Asthma Clinical Research, LLC, Oklahoma City, Oklahoma
  - Pennsylvania State University, Hershey, Pennsylvania
  - Dallas Allergy Immunology, Dallas, Texas
  - AARA Research Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - O&O Alpan, LLC, Fairfax, Virginia
  - Bellingham Asthma Allergy Clinic, Bellingham, Washington
  - The Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Subgam-VF: Subgam-VF is a 16% IgG and will be administered weekly, by subcutaneous infusion over a period of 26 weeks.
Period: Overall Study
Arm/Group | Subgam-VF
Started | 38
Completed | 33
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — withdrew consent due to AEs | 1
Not completed — Precautionary measure | 1

BASELINE CHARACTERISTICS:
Population: All subjects
Arm/Group | Subgam-VF
Number analyzed (Participants) | 38
Age, Customized [Count of Participants; unit: Participants]
  >=16 years | 25
  < 16 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Data (Derived From Absolute Concentration) Were Pooled With Historical Data and a Treatment Variable Defined (Subgam-VF or Gammaplex 5% IGIV). Outcome Measure Defined as Log Transformed sAUC0-t Standardized to One Week.
Description: Log transformed sAUC0-t, (AUC0-t standardized to one week) were analysed using a multiple linear regression model fitted including treatment, allowing for variability between treatment groups. The mean difference (Subgam-VF or Gammaplex IGIV 5%) between treatments with 90% Confidence Interval (CI) were back transformed to give an estimate of the ratio (Subgam-VF/ Gammaplex 5% IGIV) of sAUC(0-t). Data was collected at the following timepoints after week 21 of the clinical trial over a period of 1 week: Pre-dose on Day 0 and post-dose at days 1, 2, 3, 5 and 7.
Time Frame: 1 week
Population: Subgam PK Population was defined as all subjects in the ITT population who had a pre-dose sample at steady state and at least 4 post-dose samples at steady state, 1 of which should have been the Day 7 PK sample.
  Population included 50 Subjects from GMX01 (NCT00278954), 25 Subjects from GMX04 (NCT01289847) and 38 Subjects from SCIG03.
Measure: Mean (90% Confidence Interval); unit: Ratio
Groups:
- Subgam-VF and Gammaplex 5%: Subgam-VF
  Subgam-VF is a 16% IgG and will be administered weekly, by subcutaneous infusion. The total duration of treatment will be for 26 weeks.
  The initial weekly dose of Subgam-VF administered will be calculated by taking the average weekly equivalent of the subject's IGIV dose (should be stable, as in same mg/kg +/- 5%), divided by the average dosing interval in weeks (i.e. 3 or 4), multiplied by 1.37, a dose adjustment coefficient based on other licensed subcutaneous IgG products. If the subject was already receiving a weekly SCIG IgG there will be no dose adjustment.
  This population included 50 Subjects from GMX01 (NCT00278954), 25 Subjects from GMX04 (NCT01289847) and 38 Subjects from SCIG03.
Arm/Group | Subgam-VF and Gammaplex 5%
Number analyzed (Participants) | 113
Ratio | 0.98 [0.91 to 1.05]

2. Secondary Outcome: Number of Participants Who Experienced AEs Based on Treatment-emergent AEs (TEAEs)
Description: TEAEs defined as those events with onset date between the first infusion date and 28 days after the last infusion.
Time Frame: 30 weeks
Population: The intent-to-treat population included all subjects who received at least 1 infusion of Subgam-VF.
Measure: Count of Participants; unit: Participants
Groups:
- Subgam-VF: Subgam-VF is a 16% IgG and will be administered weekly, by subcutaneous infusion for a total duration of 26 weeks.
Arm/Group | Subgam-VF
Number analyzed (Participants) | 38
Participants
  Any TEAE | 36
  No TEAE | 2
  Discontinued because of TEAEs | 1
  Product Related TEAE | 15
  No Product Related TEAEs | 23
  SAE | 0

3. Secondary Outcome: Dose Refinement in Switching From Gammaplex 5% IGIV to Subgam-VF
Description: The initial weekly dose of Subgam-VF administered was calculated by taking the average weekly equivalent of the subject's IGIV dose, divided by the average dosing interval in weeks (i.e. 3 or 4), multiplied by 1.37, a dose adjustment coefficient based on other licensed subcutaneous IgG products. If the subject was already receiving a weekly SCIG IgG there will be no dose adjustment.
  A refined dose adjustment was estimated as 1.37/the ratio (Subgam-VF/ Gammaplex 5% IGIV) of geometric means for sAUC0-t and presented with 90% CI.
Time Frame: Week 26
Population: The PK Dose-Adjustment population included all those in the Subgam PK population who had previous treatment with IGIV and those in the Gammaplex 5% PK population. This population was analysed to estimate a refined dose adjustment factor.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- Subgam-VF and Gammaplex 5%: Subgam-VF is a 16% IgG and will be administered weekly, by subcutaneous infusion for a total duration of 26 weeks.
  This population included 23 Subjects from the Gammaplex PK Populations in GMX01 (NCT00278954) and 21 Subjects from GMX04 (NCT01289847), in addition included 20 Subjects from SCIG03.
Arm/Group | Subgam-VF and Gammaplex 5%
Number analyzed (Participants) | 64
Ratio | 1.33 [1.23 to 1.44]

4. Secondary Outcome: Number of Infusion Site Reactions
Description: Infusion site reactions are defined as those events with onset date between the first infusion date and 28 days after the last infusion.
Time Frame: 30 weeks
Population: Total number of participants was 38
Measure: Number; unit: infusion site reactions
Groups:
- Subgam-VF: Subgam-VF
  Subgam-VF is a 16% IgG and will be administered weekly, by subcutaneous infusion. The total duration of treatment will be for 26 weeks.
  The initial weekly dose of Subgam-VF administered will be calculated by taking the average weekly equivalent of the subject's IGIV dose (should be stable, as in same mg/kg +/- 5%), divided by the average dosing interval in weeks (i.e. 3 or 4), multiplied by 1.37, a dose adjustment coefficient based on other licensed subcutaneous IgG products. If the subject was already receiving a weekly SCIG IgG there will be no dose adjustment.
Arm/Group | Subgam-VF
Number analyzed (Participants) | 38
infusion site reactions | 447

5. Other Pre Specified Outcome: Population PK Model for IgG in PID Patients for Alternative Dosing Schedules.
Description: Develop a population pharmacokinetic (PK) model for IgG in PID patients following IV (Gammaplex 5%) or SC (Subgam-VF) administration;
  * Conduct a formal covariate analysis to assess the impact of patient demographics, and disease-related factors on the PK of IgG following IV or SC administration and to identify those patient covariates which may be utilized in or require dose adjustment;
  * Use the final population PK model to simulate serum IgG concentration-time profiles in a population of PID patients in order to:
    * Assess switching from various IgG IV and SC dosing regimens; and
    * Derive the weight-adjusted dose increment required to achieve a specified difference in serum IgG trough levels when Subgam-VF is administered either weekly or biweekly
Time Frame: 30 months
Population: The analysis population included 50 Subjects from GMX01 (NCT00278954), 25 Subjects from GMX04 (NCT01289847) and 38 Subjects from SCIG03 Clinical Trials.
  A measure type of 'number' has been used as this represents the predicted change in IgG trough levels when switching between Various IgG Dosing Regimens using a Dose Adjustment Factor of 1.37
Measure: Number; unit: % of predicted change in IgG trough
Arm/Group | Subgam-VF
Number analyzed (Participants) | 113
% of predicted change in IgG trough
  Increase from IGIV to Weekly Subgam | 31
  Increase from IGIV to Biweekly Subgam | 22
  Decrease from Weekly Subgam to Biweekly Subgam | 7
  Increase from Weekly Subgam to twice weekly Subgam | 2
  Increase from Weekly Subgam to 3x weekly Subgam | 3
  Increase from weekly Subgam to 5x weekly Subgam | 3
  Increase from weekly Subgam to 7x weekly Subgam | 3

ADVERSE EVENTS:
Time Frame: 7 months
Description: Collected during 6 months of treatment and for 28 days after the last administration of Subgam-VF
Arm/Group | Subgam-VF
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 36/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subgam-VF (N=38)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (10)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest Pain (General disorders) | 2 (2)
Fatigue (General disorders) | 3 (4)
Infusion Site Bruising (General disorders) | 2 (3)
Infusion Site Erythema (General disorders) | 6 (12)
Infusion Site Pain (General disorders) | 6 (21)
Infusion Site Pruritus (General disorders) | 4 (5)
Infusion Site Swelling (General disorders) | 2 (6)
Pain (General disorders) | 3 (5)
Pyrexia (General disorders) | 6 (11)
Acute Sinusitis (Infections and infestations) | 4 (6)
Bronchitis (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (3)
Gastroenteritis Viral (Infections and infestations) | 3 (4)
Nasopharyngitis (Infections and infestations) | 10 (15)
Pharyngitis Streptococcal (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 4 (7)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (5)
Urinary Tract Infection (Infections and infestations) | 4 (5)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 5 (6)
Ligament Sprain (Injury, poisoning and procedural complications) | 2 (2)
Tooth Fracture (Injury, poisoning and procedural complications) | 2 (2)
Coombs Direct Test Positive (Investigations) | 4 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Headache (Nervous system disorders) | 8 (12)
Haemosiderinuria (Renal and urinary disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Tooth Extraction (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT01884311/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT01884311/SAP_001.pdf